CLINICAL TRIAL: NCT00726713
Title: A 24 Week, Double-blind, Placebo-controlled, Multisite Study of Metanx® in Subjects With Type 2 Diabetic Peripheral Neuropathy (DPN)
Brief Title: Study of Metanx® in Subjects With Type 2 Diabetic Peripheral Neuropathy (DPN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamlab, Inc. (Industry)
Collaborators: Tulane University Health Sciences Center (Other); VA Nebraska Western Iowa Health Care System (U.S. Federal Agency); Scott and White Hospital & Clinic (Other); Dallas Diabetes and Endocrine Center (Other); University of Alabama at Birmingham (Other); dgd Research, Inc. (Industry); Baylor Health Care System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M-001
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-07

CONDITIONS: Type 2 Diabetic Peripheral Neuropathy (DPN)
Keywords: Metanx; diabetes; neuropathy; folic acid; folate; L-methylfolate; vitamin B6; Pyridoxal 5'-phosphate; vitamin B12; methylcobalamin
MeSH Terms: conditions — Diabetes Mellitus | interventions — metanx

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Metanx
  Interventions: Other: Metanx (a medical food)
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Metanx placebo

INTERVENTIONS:
Other: Metanx (a medical food) — Metanx one tablet twice a day
  Arms: 1
Other: Metanx placebo — Metanx placebo one tablet twice a day
  Arms: 2

SUMMARY:
The purpose of this research study is to determine if Metanx improves sensory neuropathy in persons with Type 2 diabetes. Metanx is a medical food available with a prescription from a physician. It consists of L-methylfolate, Pyridoxal 5'-phosphate, and Methylcobalamin, which are the active forms of folate, vitamin B6, and vitamin B12, respectively. Subjects will be randomly assigned to receive either Metanx or placebo for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 25 and 80 years of age (inclusive);
2. Documented diabetes mellitus Type 2 (Based upon ADA criteria);
3. Peripheral polyneuropathy: Vibration Perception Threshold (VPT) 25-45 Volts at hallux on either leg.
4. Adequate lower extremity vascular status:

   * Palpable pedal pulse in both feet;
   * No intermittent claudication;
   * No history of lower extremity vascular bypass surgery or angioplasty
5. The subject is able to understand the information in the informed consent form and is willing and able to sign the consent.

Exclusion Criteria:

1. Amputation of any kind or an ulceration within the last two (2) years including at Screen;
2. History or active Charcot neuroarthropathy on either foot;
3. Previous surgery to spine or lower extremity with residual symptoms of pain or difficulty with movement;
4. Severe rheumatoid arthritis or osteoarthritis that would cause discomfort during causal walking or stair climbing;
5. Current treatment with systemic steroids, immunosuppressives, or radiotherapy;
6. Peripheral vascular disease defined as any nonpalpable foot pulse, history of claudication, or a history of lower extremity vascular bypass surgery or angioplasty;
7. Glycated hemoglobin (HbA1c) >9 at Screen.
8. Uncontrolled heart (Hypertension: BP > 160/90), or lung disease (uncontrolled asthma or shortness of breath) in the last 2 months prior to Screen;
9. End stage kidney disorder requiring hemodialysis or serum creatinine > 2.5X (normal upper limit);
10. The following supplements within 2 months prior to Screen: alpha lipoic acid; B12 injection; >10mg of B6; or, > 800mcg of folate;
11. Taking either an opiate at any dose or on the maximum dose of any anticonvulsant;
12. Pregnant or nursing;
13. Life expectancy < 12 months;
14. Initiated therapies for Painful Diabetic Neuropathy (pregabalin, gabapentin, duloxetine etc.) in the last 2 months prior to Screen;
15. Initiated new hyperglycemic, insulin, statin or hypertensive therapies within 2 months prior to Screen (dose modifications of current therapies are allowed at the discretion of the investigator);
16. Current alcohol or drug abuse (or history of such abuse within the past 3 years); and,
17. Not willing or able to follow procedures specified by the protocol and/or the instructions of the study personnel.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Fonseca, MD, Principal Investigator — Tulane University Health Sciences Center
Locations (6):
- United States (6):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Omaha VA Medical Center, Omaha, Nebraska
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - dgd Research, Inc., San Antonio, Texas
  - Scott and White Hospital & Clinic, Temple, Texas

REFERENCES:
- [Result] Fonseca VA, Lavery LA, Thethi TK, Daoud Y, DeSouza C, Ovalle F, Denham DS, Bottiglieri T, Sheehan P, Rosenstock J. Metanx in type 2 diabetes with peripheral neuropathy: a randomized trial. Am J Med. 2013 Feb;126(2):141-9. doi: 10.1016/j.amjmed.2012.06.022. Epub 2012 Dec 5. PMID 23218892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 373 patients screened, 214 entered the study , and 200 completed. The study was conducted at 6 participating U.S. sites
Pre-assignment Details: Inclusion criteria included individuals 25 and 80 years of age, documented diabetes Type 2, Peripheral polyneuropathy, adequate lower extremity vascular status, and subject competence. 17 exclusion criteria including an HbA1c >9, uncontrolled heart or lung disease, and vitamin B supplementation, contributed to the number of screening failures.
Groups:
- Metanx: Patients aged 25 to 80 years with type 2 diabetes and neuropathy, were given Metanx (L-methylfolate calcium 3 mg, methylcobalamin 2 mg, and pyridoxal-5'-phosphate 35 mg (LMF-MC-PLP)) one tablet twice a day.
- Placebo: Patients aged 25 to 80 years with type 2 diabetes and neuropathy, were given Placebo, one tablet twice a day
Period: Overall Study
Arm/Group | Metanx | Placebo
Started | 106 | 108
Completed | 99 | 101
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Metanx: Metanx one tablet twice a day
- Placebo: Placebo one tablet twice a day
- Total: Total of all reporting groups
Arm/Group | Metanx | Placebo | Total
Number analyzed (Participants) | 106 | 108 | 214
Age Continuous [Mean (Standard Deviation); unit: years] | 62.29 (8.54) | 62.95 (9.17) | 62.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 73 | 75 | 148

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Vibration Perception Threshold (VPT) at 24 Weeks
Description: Vibration Perception Threshold (VPT) 25-45 volts at hallux on either leg as measured by VPT meter on the great toe of each foot. Mean VPT averaged across both toes.
Time Frame: VPT was measured a 0 (baseline), and 24 weeks
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
volts
  Baseline | 32.16 (13.00) | 33.88 (14.24)
  Change from Baseline Week 24 | -1.96 (13.08) | -3.27 (10.32)

2. Secondary Outcome: Change From Baseline in Neuropathy Total Symptom Score-6 (NTSS-6)
Description: This measure was taken to determine if Metanx® (compared to placebo) changes neuropathic symptoms as evaluated by the Neuropathy Total Symptom Score-6 (NTSS-6)
  The Neuropathy Total Symptom Score-6 Scale (NTSS-6) is a validated scale that evaluates individual neuropathy sensory symptoms in patients with diabetes mellitus (DM) and diabetic peripheral neuropathy (DPN). This scale was a modified 6 item scale that consists of yes or no questions. Scores range between 0 and 21.96, a higher score indicates greater severity of symptoms. After adjusting for baseline measurements scores are reflected as negative numbers. Negative numbers indicate improvement in symptoms. ie. a change from baseline after 24 weeks of -2 would be a greater improvement than a change in baseline of -1 after 24 weeks.
Time Frame: NTSS-6 scores were taken at 0 (Baseline), 16, and 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (0-6)
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
units on a scale (0-6)
  Baseline | 3.73 (1.79) | 3.45 (2.05)
  Change from Baseline Week 16 | -0.09 (1.42) | -0.40 (1.72)
  Change from Baseline Week 24 | -0.96 (1.54) | -0.53 (1.69)
Statistical Analysis 1: Comparison: Metanx vs Placebo; Change from Baseline, Week 16; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis; Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes
Statistical Analysis 2: Comparison: Metanx vs Placebo; Change from Baseline, Week 24; Test type: Superiority or Other; p = 0.033, Mixed Models Analysis; Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes

3. Secondary Outcome: Change From Baseline in Neuropathy Disability Score (NDS)at Week 16 and 24
Description: This outcome was taken to determine if Metanx® (compared to placebo) has an effect on clinical examination as determined by the Neuropathy Disability Score (NDS)
  The Neuropathy Disability Score (NDS) evaluates the severity of individual symptoms of neuropathy. A simple visual numeric distress scale is used that ranges from 0 to 10. The most favorable score is 0, which indicates an absence of symptoms. The most severe symptoms possible would be recorded as a score of 10.
Time Frame: NDS scores were taken at 0 (Baseline), 16, and 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (0-10)
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
units on a scale (0-10)
  Baseline | 7.51 (2.36) | 7.47 (2.17)
  Change from Baseline Week 16 | -0.78 (2.13) | -0.18 (2.24)
  Change from Baseline Week 24 | -0.47 (2.11) | -0.36 (2.14)
Statistical Analysis 1: Comparison: Metanx vs Placebo; Change from Baseline, Week 16; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis; Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes

4. Secondary Outcome: Change From Baseline in Plasma Marker Levels of Total Folate and Total Methyl Malonic Acid (MMA) at Week 16 and 24
Description: To determine if Metanx® (compared to placebo) affects a change in subject's total folate and total methyl malonic acid (MMA) at week 16 and 24
Time Frame: Change from Baseline in Plasma Marker Levels at 0 (Baseline), 16, and 24 weeks
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
nmol/L
  Total Folate (nmol/L) at Baseline | 42.19 (9.93) | 43.04 (9.30)
  Total Folate, Change from BL Week 16 | 7.25 (10.52) | -1.07 (8.27)
  Total Folate, Change from BL Week 24 | 7.53 (10.42) | -2.75 (8.26)
  Total methyl malonic acid (MMA) (nmol/L) at BL | 186.16 (120.11) | 195.72 (169.19)
  Total MMA, Change from BL Week 16 | -56.38 (102.72) | 13.89 (125.21)
  Total MMA, Change from BL Week 24 | -63.29 (107.00) | -15.42 (59.90)
Statistical Analysis 1: Comparison: Metanx vs Placebo; Total Folate, Change from BL, Week 16; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes
Statistical Analysis 2: Comparison: Metanx vs Placebo; Total Folate, Change from BL, Week 24; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes
Statistical Analysis 3: Comparison: Metanx vs Placebo; Total MMA, Change from Baseline Week 16; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes
Statistical Analysis 4: Comparison: Metanx vs Placebo; Total MMA, Change from BL, Week 24; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes
Statistical Analysis 5: Comparison: Metanx vs Placebo; Total Homocysteine, Change from BL, Week 16; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes
Statistical Analysis 6: Comparison: Metanx vs Placebo; Total Homocysteine, Change from BL, Week 24; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes

5. Secondary Outcome: Change From Baseline in SF-36 MCS and SF-36 PCS at Week 24
Description: To determine if Metanx® (compared to placebo) affects a subject's "quality of life" as determined by the SF-36 questionnaire
  The Short Form- 36 Mental Component Summary (SF-36 MCS) and SF-36 Physical Component Summary (SF-36 PCS) both measure health related quality of life, the MCS quantifying mental health and the PCS quantifying physical function. They are both scored on 100 point scales with 0 representing the worst possible outcome and 100 representing the most optimal possible scoring
Time Frame: SF-36 MCS and SF-36 PCS scores were measured at 0 (Baseline) and 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (0-100)
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
units on a scale (0-100)
  SF-36 PCS, Baseline | 40.74 (10.30) | 39.03 (9.81)
  SF-36 PCS, Change from BL, Week 24 | 0.03 (8.34) | 0.87 (8.21)
  SF-36 MCS, Baseline | 50.96 (9.87) | 52.66 (8.39)
  SF-36 MCS, Change from BL, Week 24 | 1.99 (8.57) | -0.29 (8.48)
Statistical Analysis 1: Comparison: Metanx vs Placebo; SF-36 MCS, Change from BL, Week 24; Test type: Superiority or Other; p = 0.0306, Mixed Models Analysis — Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes

6. Secondary Outcome: Change From Baseline in 10-point Visual Analog Scale(VAS) at Week 24
Description: To determine if Metanx® (compared to placebo) affects a subject's lower extremity pain level using a 10-point Visual Analog Scale at Baseline and 24-week evaluation visits.
  The Visual Analog Scale (VAS) measures a patients sensation of pain. A 10-cm visual analog scale is used. A measurement on the 10 cm analog scale is used to quantify the level of pain indicated with 0 cm indicating "no pain" and 10 cm indicating the "worst pain imaginable".
Time Frame: VAS scores were taken at 0 (Baseline) and 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (0-10)
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
units on a scale (0-10)
  VAS Baseline | 3.26 (2.77) | 3.25 (2.76)
  VAS, Change from BL, Week 24 | -0.27 (2.28) | -0.03 (2.61)

7. Secondary Outcome: (Exploratory) Change From Baseline in Levels of IL-6 and TNF-α, at Week 24
Description: (Exploratory) To determine if Metanx® affects a subject's plasma oxidative stress and inflammatory marker levels, including IL-6 and TNF-α
Time Frame: Analyte levels were taken at 0 (Baseline) and 24 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
pg/mL
  IL-6 (pg/mL), Baseline | 3.66 (2.91) | 3.68 (3.01)
  IL-6, Change from BL, Week 24 | -0.25 (2.60) | 0.07 (2.42)
  TNF-a (pg/mL), Baseline | 1.69 (1.25) | 2.01 (2.72)
  TNF-a, Change from BL, Week 24 | 0.03 (0.76) | -0.04 (0.54)

8. Secondary Outcome: (Exploratory) Change From Baseline in the Hospital Anxiety and Depression Scale (HADS) Question Inventory at Week 24
Description: The Hospital Anxiety and Depression Scale (HADS) consists of a 14-item questionnaire that provides a measurement of depression. Each item is rated on a 4-point scale, giving a maximum scores of 21 for the most severe depression. Depression was evaluated using the Hospital Anxiety and Depression Scale (HADS) question inventory at Baseline, and 24-week evaluation visits
Time Frame: HADS Scores scores were taken at 0 (Baseline) and 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (0-21)
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
units on a scale (0-21)
  HADS Depression, Baseline | 4.16 (3.24) | 4.42 (3.12)
  HADS Depression, Change from BL, Week 24 | -1.03 (2.53) | -0.45 (2.58)
Statistical Analysis 1: Comparison: Metanx vs Placebo; HADS Depression, Change from BL, Week 24; Test type: Superiority or Other; p = 0.054, Mixed Models Analysis; Generalized linear mixed models were used to assess baseline for continuous and discrete outcomes

9. Secondary Outcome: Change From Baseline in Total Homocysteine at Week 16 and 24
Description: To determine if Metanx® (compared to placebo) affects change in subjects total homocysteine levels
Time Frame: Change from Baseline in Plasma Marker Levels at 0 (Baseline), 16, and 24 weeks
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
µmol/L
  Total homocysteine (µmol/L) at Baseline | 9.71 (4.29) | 9.47 (3.90)
  Total homocysteine, Change from BL Week 16 | -2.70 (2.90) | 0.58 (2.58)
  Total homocysteine, Change from BL Week 24 | -2.68 (2.98) | 0.48 (2.40)

10. Secondary Outcome: (Exploratory) Change From Baseline in Levels of Hs-CRP at Week 24
Description: (Exploratory) To determine if Metanx® affects a subject's plasma oxidative stress and inflammatory markers levels including hs-CRP
Time Frame: Analyte levels were taken at 0 (Baseline) and 24 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
mg/L
  hs-CRP (mg/L), Baseline | 6.46 (5.98) | 7.44 (7.23)
  hs-CRP, Change from BL, Week 24 | -0.71 (4.05) | 0.13 (4.15)

11. Secondary Outcome: (Exploratory) Change From Baseline in Levels Potential Antioxidant (PAO) at Week 24
Description: (Exploratory) To determine if Metanx® affects a subject's plasma oxidative stress and inflammatory markers levels including Potential Antioxidant (PAO)
Time Frame: Analyte levels were taken at 0 (Baseline) and 24 weeks
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Metanx | Placebo
Number analyzed (Participants) | 106 | 108
µmol/L
  PAO (µmol/L), Baseline | 1094.52 (230.83) | 1102.15 (250.54)
  PAO, Change from BL, Week 24 | 7.95 (190.36) | 5.29 (204.92)

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) included events starting on or after the baseline visit until 4 weeks after the last study visit on week 24. The total duration of AE monitoring was 196 days.
Description: An adverse event is any undesirable sign, symptom or medical condition occurring after starting study drug, even if the event is not considered to be related to study drug.
  Adverse Event reporting was provided only with specificity to the affected Organ System. Additional detail was not available at the time of reporting.
Arm/Group | Metanx | Placebo
Serious Adverse Events (participants affected / at risk) | 5/106 | 8/108
Other Adverse Events (participants affected / at risk) | 25/106 | 27/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metanx (N=106) | Placebo (N=108)
Transient Ischemic Attack (Vascular disorders) | 2 (2) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Ligament Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary Artery Bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Cardiac Failure, Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metanx (N=106) | Placebo (N=108)
Infections and infestations (Infections and infestations) | 6 (6) | 6 (6)
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
General disorders and administration site conditions (General disorders) | 4 (4) | 3 (3)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Surgical and medical procedures (Surgical and medical procedures) | 3 (3) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Adverse Event reporting detailed in the "Other Adverse Events" section was provided only with specificity to the affected Organ System. Additional detail for the "Other Adverse Events" was not available at the time of reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay publication of study results until after multi-center results were published or, a period of up to 20 months had elapsed after termination of the study, whichever shall occur first.